CLINICAL TRIAL: NCT04125446
Title: Genomic and Epigenomic Alterations After Cancer Treatment in Pregnancy
Acronym: GE-CIP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Gasthuisberg (Other)
Collaborators: University Hospital, Antwerp (Other); University Hospital, Ghent (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Frederic Amant, Clinical Professor, Principal Investigator, University Hospital, Gasthuisberg
Other Study IDs: S62388
Record Dates: First submitted 2019-10-10; First posted 2019-10-14 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Cancer; Pregnancy
Keywords: cancer in pregnancy; chemotherapy; offspring; genotoxicity
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Biospecimen Retention: Samples With DNA — Parental blood, cord blood, meconium, buccal swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cancer in pregnancy chemo treated: Patients that received at least one of the following treatments: Carboplatin, Cisplatin, Cyclophosphamide, Paclitaxel and/or anthracyclines, the latter being the most given type of CT during pregnancy
- Cancer in Pregnancy not chemo treated: Women who were not treated with CT during pregnancy, including those who were solely surgically treated or did not receive any treatment during pregnancy, will be included in the CT-unexposed control arm
- healthy pregnancies: A group of healthy pregnant women without cancer will form the second control group

SUMMARY:
The investigators want to obtain a fundamental understanding if and which chemotherapeutic agents used for treating cancer during pregnancy are associated with placental and/or offspring (epi)genetic changes, potentially causing FGR and childhood/adult diseases later in life.

DETAILED DESCRIPTION:
Rationale: Cancer is the second leading cause of death during the reproductive years and affects between 1:1000 and 2000 pregnant women. Previous studies from our group have shown that chemotherapeutic cancer treatment in pregnancy has reassuring outcomes in terms of cognitive and cardiac neonatal outcomes, and hence has been proposed as standard of care. However fetal growth restriction (FGR), which places an infant at significant risk of perinatal morbidity and mortality, is more common in women who were systemically treated during pregnancy compared to the non-cancer population. The possibility that chemotherapy during pregnancy causes placental (epi)genetic damage, and consequently induces FGR, or affects offspring DNA leading to potential deleterious effects later in life, such as cancer or other diseases, has not been investigated so far. As the cytotoxic effects of chemotherapy at DNA level have been well established, it could be speculated that chemotherapy-induced DNA damage may interfere with fetal and childhood health in the long term. The results of this study will lead to an increased understanding of potential toxic effects of chemotherapy for the unborn child and may therefore contribute to the development of safe and solid treatment regimens for pregnant cancer patients and their children.

Objectives: To obtain a fundamental understanding if and which chemotherapeutic agents used for treating cancer during pregnancy are associated with offspring (epi)genetic changes, potentially causing FGR and childhood/adult diseases later in life.

Study design: This international multicentre prospective observational trial functions as an extension of the CIP-study (Cancer in Pregnancy, S25470) and aims to collect cord blood, meconium and neonatal buccal cells at birth. Parental peripheral blood and buccal cells will be collected and used as reference. Minimal requirement to participate in this study is participation in Part I.IA of the original CIP-study. Through this CIP-study we are able to gather pregnancy-, malignancy- and placenta-related data.

Study population: All patients with histological proven cancer during pregnancy and an ongoing pregnancy (≥24 weeks of gestation) treated with chemotherapy (alkylating agents, anthracyclines, taxanes and/or platinum derivates) or other treatment options (surgery, radiotherapy and/orsystemic treatment other than chemotherapy, or none).

Main study parameters/endpoints: determination of potential (epi)genetic alterations in cord bloodand buccal cells of the newborn, and the association with chemotherapy concentrations measured in newborn tissue.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: There are no risks associated nor benefits expected with participation in this study.

ELIGIBILITY:
Inclusion Criteria:

* Cancer in pregnancy - CT-treated arm

  * Histological proven cancer during pregnancy (any type and stage)
  * (Former) participation in part I.IA of the CIP-study S25470 (and I.IB for the placental sub study)
  * Treatment during pregnancy with one or a combination of the following chemotherapeutic agents:
* Cyclophosphamide
* Anthracyclines
* Taxanes
* Platinum derivates

  * Gestational age (GA) at birth ≥24 weeks Cancer in pregnancy - CT-untreated arm
  * No treatment during pregnancy or surgery only (subgroup 1)
  * Radiotherapy and/or systemic treatment (other than CT) during pregnancy (subgroup 2)
  * GA at birth ≥24 weeks Healthy pregnant controls
  * matched for maternal age, gestation at birth and infant gender with CT-treated arm
  * GA at birth ≥24 weeks (only for placental study)

Exclusion Criteria:

* GA at birth <24 weeks (miscarriage or termination of pregnancy) (placental study)
* Mentally disabled women or patients who have a significantly altered mental status that would prohibit the understanding and giving of informed consent
* Any comorbidity that is associated with an enhanced risk of placental pathology or FGR such as hypertensive disorders, preeclampsia, (gestational) diabetes, SLE, Crohn's disease, renal or cardiac pathology (healthy pregnant controls)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The current study will focus on patients that received at least one of the following treatments: carboplatin, cisplatin, cyclophosphamide, paclitaxel and/or anthracyclines, the latter being the most given type of CT during pregnancy (cfr. also Table 1). Women who were not treated with CT during pregnancy, including those who were solely surgically treated or did not receive any treatment during pregnancy, will be included in the CT-unexposed control arm.In the CT-unexposed arm, we will also include women that had systemic treatment other than chemotherapy (e.g. targeted therapies) and/or radiotherapy. A group of healthy pregnant women without cancer, delivering in our participating centres, will form the second control group.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-10-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessing general genotoxicity of fetal DNA; genomic instability, de novo somatic mutations and methylation changes related to in utero exposure to chemotherapy | through study completion, an average of 5 years
  somatic mutations, structural alterations, methylation changes

SECONDARY OUTCOMES:
Measuring concentration of chemotherapeutic drugs in offspring tissue (cord blood, meconium) in patients receiving cisplatin, carboplatin and/or cyclophosphamide treatment. | through study completion, an average of 5 years
  DNA adduct

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Amant, MD,PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium